CLINICAL TRIAL: NCT05444699
Title: Oral Prednisolone for Acute Rhinovirus Induced Wheezing in Children Less Than 2 Years of Age: a Point-of-care Testing Guided Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Oral Prednisolone for Acute Rhinovirus Induced Wheezing in Children Less Than 2 Years of Age
Acronym: RhinoPOCRCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Terhi Tapiainen, Professor of Pediatrics, Head of Pediatric Infectious Diseases and Emergency Department, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OY102021; 2024-512561-13-00 (EU CTIS Number); 2021-006050-31 (EudraCT Number)
Record Dates: First submitted 2021-12-22; First posted 2022-07-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Bronchiolitis Acute Viral
MeSH Terms: interventions — prednisolone phosphate; High Fructose Corn Syrup

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone (Experimental): Prednisolone Sodium Phosphate (25 mg/5 mL) oral suspension administered 1 mg/kg* (up to 20 mg = 4 mL) once a day for 3 days.
  *(0-5 kg: 5 mg; 5.01-7.5 kg: 7.5 mg; 7.51-10 kg: 10 mg; 10.01-12.5 kg: 12.5 mg; 12.51-15 kg: 15 mg; 15.01-17.5 kg: 17.5 mg; ≥ 17.51 kg: 20 mg)
  Interventions: Drug: Prednisolone Sodium Phosphate
- Placebo (Placebo Comparator): Sugar syrup oral suspension containing saccharum 630-640 mg/g and aqua purificata 360-370 mg/g administered the same amount in milliliters as experimental product (up to 4 mL) once a day for 3 days.
  Interventions: Drug: Sugar syrup

INTERVENTIONS:
Drug: Prednisolone Sodium Phosphate — Oral suspension administered 1 mg/kg once a day for three days
  Arms: Prednisolone
Drug: Sugar syrup — Oral suspension administered the same amount in milliliters as experimental product once a day for three days
  Arms: Placebo

SUMMARY:
The aim of the trial is to evaluate whether the use of oral prednisolone directed by point-of-care testing is useful in acute wheezing caused by rhinovirus in children aged 6-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Wheezing bronchitis diagnosed by a physician
* Need for salbutamol treatment at the emergency department
* Positive nasopharyngeal rhinovirus or picornavirus finding in point-of-care testing

Exclusion Criteria:

* Need for immediate resuscitation
* Immediate transfer to ICU
* Suspected pneumonia based on the auscultation finding
* Suspected serious bacterial infection
* Other respiratory virus finding in the absence of rhinovirus or picornavirus
* Positive respiratory syncytial virus finding
* Positive SARS-coronavirus-2 finding
* Positive Mycoplasma pneumoniae finding
* Positive Bordetella pertussis finding
* Contact with a person with chickenpox within 14 days
* Active chickenpox
* Suspected foreign body of the respiratory tract
* Immunosuppressive treatment
* Systemic corticosteroid treatment within 14 days
* Allergy to corticosteroids

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Within 7 days of study entry
  The difference (in minutes) between the study entry and the time that the patient is deemed to be fit for discharge (sign off for discharge)
  Subgroup analyses for the primary outcome are performed in following subgroups:
  * Children presenting with first episode of wheezing
  * Children with at least one previous episode of wheezing diagnosed by a physician
  * Children with a cycle threshold number of < 30 for detected picornavirus
  * Children with a cycle threshold number of 30-37 for detected picornavirus
  * Children with a cycle threshold number of 38-40 for detected picornavirus

SECONDARY OUTCOMES:
Total length of hospital stay | Within 7 days of study entry
  The difference (in minutes) between the study entry and the actual time of discharge from the hospital
Intensive care unit (ICU) admissions | Within 7 days of study entry
  Proportion of children admitted to ICU
Supplemental oxygen | Within 7 days of study entry
  The total duration (in minutes) of the need for supplemental oxygen
Pediatric Early Warning Signs (PEWS) score | Within 7 days of study entry
  Maximum decrease in PEWS score within 12 hours after study entry. PEWS scores range from 0 to 32 depending on the child's respiratory rate, work of breathing, saturation of peripheral oxygen, need for supplemental oxygen, blood pressure, heart rate, capillary refill and level of consciousness. 0 refers to low and > 7 to high risk of deterioration.
Recurrence of wheezing | Within 56 days of study entry
  Proportion of patients with recurrence of wheezing after initial episode
Hospital re-admission | Within 14 days of study entry
  Proportion of patients with re-admission to hospital or visit to emergency department after discharge from the hospital
Proportion of patients with cough at 14 days of study entry | At 14 days of study entry
  Proportion of patients with cough at 14 days of study entry
Duration of cough | Within 28 days of study entry
  Mean duration (in days) of cough without relapse for 3 days
Duration of cough | Within 14 days of study entry
  Mean duration (in days) of cough without relapse for 3 days
Duration of salbutamol use | Within 14 days of study entry
  Mean number of days in which salbutamol is used
Duration of respiratory distress | Within 14 days of study entry
  Mean duration (in days) of respiratory distress without relapse for 3 days
Deaths | Within 30 of study entry
  Proportion of patients who died of any cause
Recurrence of wheezing (proportion) | Within 12 months of study entry
  Proportion of patients with recurrence of wheezing diagnosed by a physician at 2 and 12 months of study entry
Recurrence of wheezing (time) | Within 12 months of study entry
  Time (in days) to recurrence of wheezing diagnosed by a physician
Daily administrated asthma medication | Within 24 months of study entry
  Time (in days) to prescription of daily administrated asthma medication
Antibiotics and asthma medications | Within 24 months of study entry
  Purchases of antibiotics and asthma medications

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - SOITE Lastenpäivystys, Kokkola
  - OYS Lastenpäivystys, Oulu

IPD SHARING:
Plan to Share IPD: No